CLINICAL TRIAL: NCT01055808
Title: A Prospective, Non-safety Observational Study in Japanese Type 2 Diabetes Patients(INSIGHTS)
Brief Title: Observational Study in Japanese Type 2 Diabetes Patients
Acronym: INSIGHTS
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Other Study IDs: 13614; F3Z-JE-PV06 (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-01-23; First posted 2010-01-26 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Insulin; ITR-QOL; DTSQ; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulins

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 diabetes treated with insulin
  Interventions: Drug: Insulins

INTERVENTIONS:
Drug: Insulins — Individual dose and frequency and duration as determined by the treating physician

SUMMARY:
This study is designed to address the gap in the literature related to changing treatment regimen or formulation between different types of insulin, and how this change impacts quality of life, adherence, individual patient treatment satisfaction and glycemic control.

DETAILED DESCRIPTION:
To measure changes in Health Related Quality of Life (as measured by the Insulin Therapy Related-Quality of Life: ITR-QOL) in insulin treated type 2 diabetes over a 12 weeks period following a significant change in insulin treatment regimen. Definition of significant change is a) increase or decrease the in number of injections per day, or/and b) change in formulation of insulin (human or analog insulin, basal or bolus, rapid or mix insulin), and/or c) change in administration method (syringe or pen, disposal or re-usable).

ELIGIBILITY:
Inclusion Criteria:

* Inpatients or outpatients with type 2 diabetes, aged 20 years or older, on insulin therapy who have planned to change insulin therapy during the registration period of the study
* Patients who have provided written informed consent to participation in the study after receiving explanations about the objective and other details of the study
* Patients who have received the same insulin therapy for 3 months or longer before informed consent. (i.e. receiving the same type of insulin preparation at the same dosing frequency regardless of insulin dose)

Exclusion Criteria:

* Patients who have planned to discontinue insulin therapy
* Patients incapable of completing the ITR-QOL, DTSQ and patient's questionnaire based on their self-ratings
* Patients with type 1 diabetes
* Patients who have used CSII or have planned to switch to CSII(continuous subcutaneous insulin infusion )
* Patients with poor treatment compliance as determined by their investigators based on the treatment history

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Japanese patients with type 2 diabetes who are treated with insulin and about to have significant treatment change.
Sampling Method: Probability Sample
Enrollment: 677 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Changes in Health Related Quality of Life (ITR-QOL) in insulin treated type 2 diabetes at baseline and 12 weeks after a significant change in insulin treatment regimen | Baseline, 12 weeks

SECONDARY OUTCOMES:
Summarize by occurrence the reason for insulin treatment change at study entry | Baseline
Change in HbA1c at baseline and 12 weeks after a significant change in insulin treatment regimen | Baseline, 12 weeks
Change in treatment adherence at baseline and 12 weeks after a significant change in insulin treatment regimen | Baseline, 12 weeks
Change in DTSQ (Diabetes treatment satisfaction questionnaire) at baseline and 12 weeks after a significant change in insulin treatment regimen | Baseline, 12 weeks
Total daily dose of insulin | Baseline, over 12 weeks
Change in type of insulin product | Baseline, 12 weeks
Change from baseline in use of concomitant oral hypoglycemic drugs | Baseline, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri from 9AM-5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo, Japan

REFERENCES:
- [Derived] Ishii H, Terauchi Y, Jinnouchi H, Taketsuna M, Takeuchi M, Imaoka T. Effects of insulin changes on quality of life and glycemic control in Japanese patients with type 2 diabetes mellitus: The insulin-changing study intending to gain patients' insights into insulin treatment with patient-reported health outcomes in actual clinical treatments (INSIGHTs) study. J Diabetes Investig. 2013 Nov 27;4(6):560-70. doi: 10.1111/jdi.12086. Epub 2013 Apr 30. PMID 24843710